CLINICAL TRIAL: NCT00339248
Title: Risk of Breast Cancer and Hyperplastic Conditions in the Breast Cancer Serum Bank in Relation to Inherited Genetic Variants
Brief Title: Markers for Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905061; 05-C-N061; NCT00898586 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2007-10

CONDITIONS: Breast Cancer
Keywords: Hyperplasia; Atypia; Polymorphism; Progression; Epidemiology
MeSH Terms: conditions — Breast Neoplasms; Hyperplasia; Disease Progression

SUMMARY:
This study will analyze blood samples to identify substances that are associated with the development of breast cancer. It will determine if:

* Women who are diagnosed with a benign breast condition that is related to a considerably increased risk of breast cancer are more likely to have certain gene variants than women diagnosed with conditions related to very little increased breast cancer risk
* Women with benign breast conditions who subsequently develop breast cancer are more likely to have certain gene variants than women with similar benign conditions who do not develop breast cancer.

This study will examine blood samples from premenopausal women who underwent breast biopsy (removal of a small piece of breast tissue for microscopic examination) at four hospitals in Grand Rapids, MI, from 1977 to 1987 and were found to have benign breast disease. The women, who agreed to participate in a study of markers for breast cancer, also provided a blood sample and were interviewed for information on their breast cancer risk factors, family history of breast cancer, use of medications, and history of medical conditions.

This study will retrieve the biopsy reports for these women, determine which of them later developed breast cancer, and perform genotyping on their blood samples.

The information from this study may help in future diagnosis and treatment of breast cancer.

DETAILED DESCRIPTION:
Prevention and treatment of intraepithelial neoplasia and benign pre-malignant conditions has become an important focus of the NCI's 2015 goal of eliminating suffering and death due to cancer, although very little is known about the factors that influence development of frank malignancy in those with high risk benign/precursor conditions. The Radiation Epidemiology and Biostatistics Branches of the NCI propose to evaluate the contribution of inherited genetic variation to benign pre-malignant breast conditions, and to subsequent breast cancer risk in women diagnosed with such conditions, in the Breast Cancer Serum Bank, a unique biospecimen resource housed at NCI since 1995. Premenopausal participants (N=2632) biopsied at an average age of 27 in 1977-1987, (many diagnosed with high risk benign breast conditions (moderate/florid breast hyperplasia and atypia)) were interviewed and provided a blood sample. Participant biopsy reports will be obtained for review and recoding, and participants will be traced for vital status and breast cancer development (expected n = 240 cases). Variants in genes related to hormone metabolism and cell signaling, processes implicated in the development of premalignant breast conditions, and in genes associated with cell cycle control and apoptosis, and thus possibly related to progression to breast cancer among women with premalignant breast conditions will be assessed at the NCI Central Genotyping Facility. We have a remarkable opportunity in this study to address scientific questions regarding breast carcinogenesis mechanisms at relatively little cost. Greater comprehension of the influence of inherited factors on distinct steps in the biological pathway, first from normal tissue to benign high risk breast tumors, and then hence the breast cancer, should contribute to our understanding of the molecular mechanisms that shape breast cancer development, and holds promise for the discovery and delivery of sound risk-adapted interventions for women with high risk premalignant conditions.

ELIGIBILITY:
* INCLUSION/EXCLUSION CRITERIA:

Potentially eligible premenopausal women include 2636 who did not have a previous or concurrent (within 60 days) diagnosis of breast cancer at the time of initial benign breast biopsy (study entry) and who have at least 4 mls of serum stored in the Frederick biorepository.

Of those 2636, four women have a code indicating "refused study" in the "follow-up" variable, and despite evidence of their consent to the original study, will be omitted from all future use of study data or specimens.

Participants also will be required to be Caucasian or African American (2599 or 98.6%), and to have a pathology report successfully retrieved from a participating hospital for review.

All sample sizes subsequently cited in the text take these inclusion criteria into account, and those cited for objective 2 also incorporate adjustment for loss to follow-up.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2632
Dates: Start 2004-12

CONTACTS AND LOCATIONS:
Locations (1):
- NCI Frederick Cancer Research Center, Frederick, Maryland, United States

REFERENCES:
- [Background] Alle KM, Henshall SM, Field AS, Sutherland RL. Cyclin D1 protein is overexpressed in hyperplasia and intraductal carcinoma of the breast. Clin Cancer Res. 1998 Apr;4(4):847-54. PMID 9563877
- [Background] Blomeke B, Bennett WP, Harris CC, Shields PG. Serum, plasma and paraffin-embedded tissues as sources of DNA for studying cancer susceptibility genes. Carcinogenesis. 1997 Jun;18(6):1271-5. doi: 10.1093/carcin/18.6.1271. PMID 9214613
- [Background] Boyd NF, Jensen HM, Cooke G, Han HL. Relationship between mammographic and histological risk factors for breast cancer. J Natl Cancer Inst. 1992 Aug 5;84(15):1170-9. doi: 10.1093/jnci/84.15.1170. PMID 1635085